CLINICAL TRIAL: NCT00390585
Title: Prospective, Randomized, Comparative Study to Evaluate the Effect of Iodixanol 320 Compared to Iomeprol 350 on Contrast Medium Induced Nephropathy in Patients With Impaired Renal Function Undergoing PCI
Brief Title: Iodixanol vs. Iomeprol to Prevent Contrast-Induced Nephropathy After Coronary Intervention (CONTRAST)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GE IDE No. E00605
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2010-03-15 (Estimated); Status verified 2008-02

CONDITIONS: Renal Insufficiency, Chronic; Angioplasty, Transluminal, Percutaneous Coronary; Coronary Arteriosclerosis
Keywords: Renal Insufficiency; Angioplasty, Transluminal, Percutaneous Coronary; Contrast media
MeSH Terms: conditions — Renal Insufficiency, Chronic; Coronary Artery Disease; Renal Insufficiency | interventions — iodixanol; iomeprol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Iodixanol 320
  Interventions: Drug: Iodixanol 320
- B (Active Comparator): Iomeprol 350
  Interventions: Drug: Iomeprol 350

INTERVENTIONS:
Drug: Iodixanol 320 — Iodixanol 320 is used as contrast media while coronary intervention.
  Other Names: VISIPAQUE (TM)
  Arms: A
Drug: Iomeprol 350 — Iomeprol 350 is used as contrast media while coronary intervention.
  Other Names: Imeron
  Arms: B

SUMMARY:
The purpose of this study is to demonstrate that Iodixanol 320 is associated with a lower incidence of contrast-induced nephropathy (CIN) when compared with hyperosmolar contrast medium Iomeprol 350 in patients with impaired renal function undergoing percutaneous coronary interventions (PCI).

DETAILED DESCRIPTION:
Iodixanol, an iso-osmolar, dimeric, non-ionic contrast agent has been shown to reduce the risk of developing CIN in patients with elevated serum creatinine concentrations compared to low-osmolar contrast agents. However, no information is available about a potential protective effect of Iodixanol in patients with impaired renal function on CIN when used during PCI. Due to the high volume of contrast exposition, patients with impaired renal function are at increased risk for the development of CIN compared to patients with normal excretory renal function.

The purpose of the investigation is to determine the changes of renal function in patients with impaired renal function receiving Iodixanol 320 or Iomeprol 350 for percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal failure
* Informed, written consent

Exclusion Criteria:

* Cardiogenic shock
* Dialysis
* kidney transplantation
* Concurrent intake of nephrotoxic medication
* Planned or proceeded parenteral (i.v. or i.a.) administration of iodine-containing contrast medium at least 7 days before/after catheterization.
* Contra-indications for the use of Iodixanol (e.g. allergies)
* Women who are known to be pregnant, who are of childbearing potential and test positive for pregnancy, who have given birth within the last 90 days, who are breastfeeding
* Patient's inability to fully cooperate with the study protocol.
* Previous enrollment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2006-07; Primary Completion 2008-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Contrast-induced nephropathy after percutaneous coronary intervention during primary hospitalization | primary hospitalization

SECONDARY OUTCOMES:
Duration of primary hospitalization | Duration of primary hospitalization
Incidence of severe acute kidney failure | severe acute kidney failure
Contrast-induced nephropathy six months after PCI | 6 months
Mortality and myocardial infarction at 6 and 12 months | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schoemig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Rainer Wessely, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - 1. Medizinische Klinik, Klinikum rechts der Isar, München

REFERENCES:
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. Diabet Med. 1998 Jul;15(7):539-53. doi: 10.1002/(SICI)1096-9136(199807)15:73.0.CO;2-S. PMID 9686693
- [Result] Wessely R, Koppara T, Bradaric C, Vorpahl M, Braun S, Schulz S, Mehilli J, Schomig A, Kastrati A; Contrast Media and Nephrotoxicity Following Coronary Revascularization by Angioplasty Trial Investigators. Choice of contrast medium in patients with impaired renal function undergoing percutaneous coronary intervention. Circ Cardiovasc Interv. 2009 Oct;2(5):430-7. doi: 10.1161/CIRCINTERVENTIONS.109.874933. Epub 2009 Sep 22. PMID 20031753